CLINICAL TRIAL: NCT05657379
Title: The Effect of Product X Moisturizer on Skin Texture of Middle-Aged Women in Malaysia
Brief Title: Effect of Moisturizer on Malaysian Women Facial Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RMC/EC41/2022
Record Dates: First submitted 2022-12-07; First posted 2022-12-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Middle-aged women, moisturizer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Product X moisturizer (Experimental): Participants will used Product X moisturizer twice daily for 8 weeks
  Interventions: Other: Other: Product X moisturizer

INTERVENTIONS:
Other: Other: Product X moisturizer — Product X moisturizer containing Hyaluronic Acid and Rosa Damascena Flower Water

SUMMARY:
The goal of this clinical trial is to evaluate the effect of Product X on facial skin of middle-aged women in Malaysia. The main questions it aims to answer are:

1. The effect of Product X on skin hydration of middle-aged women in Malaysia.
2. The effect of Product X on skin elasticity of middle-aged women in Malaysia.
3. The effect of Product X on skin wrinkle of middle-aged women in Malaysia.
4. To observe any adverse effect occurrence with the use of Product X.

Participants will used Product X for 8 week and the skin assessment will be carried out at baseline, week 2, 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Middle-aged woman (40-60 years old)

Exclusion Criteria:

* Participants taking isotretinoin
* Immunocompromised patients or participants with any skin diseases or diseases that may compromised the participants well-being and study outcome.
* Participant who undergo any cosmetic procedures such as laser & light treatment for the past three months.
* Participant with a history of facial surgery.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration from baseline and at week 2, 4 and 8 after using Product X | Baseline, week 2, 4 and 8
  Skin hydration will be assessed using JANUS III skin analyzer
Change in skin elasticity from baseline and at week 2, 4 and 8 after using Product X | Baseline, week 2, 4 and 8
  Skin elasticity will be assessed using JANUS III skin analyzer
Change in skin wrinkles from baseline and at week 2, 4 and 8 after using Product X | Baseline, week 2, 4 and 8
  Skin wrinkles will be assessed using JANUS III skin analyzer and Wrinkle Severity Rating Scale (WSRS). For WSRS, dermatologists will evaluate participants' wrinkles based on 5-point photonumeric rating scale that will objectively evaluate the severity of crow's feet at rest (static) and with a smiling expression (dynamic). The scale scores are 0 for no wrinkles, 1 for very fine wrinkles, 2 for fine wrinkles, 3 for moderate wrinkles, and 4 for severe wrinkles.
Adverse effect after using Product X | Week 8
  Based on adverse effect occurrence on participants that occur during study period (8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No